CLINICAL TRIAL: NCT02386956
Title: Evaluation of Hamstrings Elongation After Different Physiotherapy Stretching Techniques
Brief Title: Hamstring Stretch Effect (STRETCH-HAMS)
Acronym: STRETCH-HAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Carlos Lozano Quijada, PT, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPC.CLQ.01.15
Record Dates: First submitted 2015-03-07; First posted 2015-03-12 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-06

CONDITIONS: Postural; Defect
Keywords: manual therapy; muscle chains; Dynamic stretching; Active stretching
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active stretching (Experimental): 10 minutes of Postural Global Reeducation for the posterior muscle chain
  Interventions: Other: Active stretching
- Dynamic Stretching (Experimental): 10 minutes of sciatic nerve manual movilization in two legs
  Interventions: Other: Dynamic Stretching
- Control (Placebo Comparator): 10 minutes with the patient lying on a machine off of magnetotherapy
  Interventions: Other: Control

INTERVENTIONS:
Other: Active stretching — 10 minutes of active stretching of the posterior muscle chain with RPG techniques
  Other Names: Postural Global Reeducation
  Arms: Active stretching
Other: Dynamic Stretching — 10 minutes of dynamic stretching of the sciatic nerve and the posterior muscle chain with manual techniques of mobilization the nerves
  Other Names: Mobilization of sciatic nerve
  Arms: Dynamic Stretching
Other: Control — 10 minutes with the patient lying on a machine off of magnetotherapy
  Other Names: Placebo
  Arms: Control

SUMMARY:
Randomized clinical trial to evaluate the elongation of the hamstrings after making different types of stretching. One group receives a stretch of global postural reeducation (RPG), another group receives a mobilization of sciatic nerve, and a third group received a placebo treatment. The evaluation of these treatments are done previously, immediately after and 20 min later. The test used to evaluate elongation are the Sit and Reach and active knee extension (AKE test).

DETAILED DESCRIPTION:
Randomized clinical trial to evaluate the elongation of the hamstrings after making different types of stretching and mobilizations used in physiotherapy. This study is realized with university students to be long time studying in sitting position, and each subject is randomly assigned to one of three different groups. One group receives 10 minutes of global postural reeducation stretching (RPG), another group receives 10 minutes of bilateral mobilization of sciatic nerve, and a third group received a placebo treatment. The evaluation of these treatments are done previously, immediately after and 20 min later. The test used to evaluate elongation are the Sit and Reach and active knee extension (AKE test). The order of measurement of each test is also randomized in each subject. The intervention is always applied to the same physical therapist, and measurements were always performed by another physiotherapist blinded.

ELIGIBILITY:
Inclusion Criteria:

* college students spend four hours or more for day sitting

Exclusion Criteria:

* college students do not spend four hours or more for day sitting
* subjects with a traumatic problem, injuries or subjects in treatment of this injuries at the moment of the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Sit and Reach test | 3 minutes
  This test involves sitting on the floor with legs out straight ahead. Feet (shoes off) are placed with the soles flat against the box, shoulder-width apart. Both knees are held flat against the floor by the tester, if required. With hands on top of each other and palms facing down, the subject reaches forward along the measuring line as far as possible. After three practice reaches, the fourth reach is held for at least two seconds while the distance is recorded. Make sure there are no jerky movements, and that the fingertips remain level and the legs flat. he score is recorded to the nearest centimeter or half inch as the distance reached by the tip of the fingers.
AKE Test | 3 minutes
  Participants were assessed on a plinth in the supine position with both lower extremities extended. Both anterior superior iliac spines were positioned by aligning them with the vertical bars of the apparatus. The lower extremity not being measured was secured to the plinth using a strap across the lower third of the thigh. Each assessor marked the lateral knee joint line with washable ink. The participants were told to flex the hip until the thigh touched the horizontal metalic bar. While maintaining the contact between the thigh and horizontal bar, the participants were asked to extend the leg as much as possible while keeping their foot relaxed and to hold the position for about 5 seconds. A standard universal goniometer was placed over the previously marked joint axis, and the inclinometer arms were aligned along the femur and fibula.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Lozano-Quijada, MPT, Principal Investigator — Universidad Miguel Hernandez de Elche; Emilio J Poveda-Pagán, PhD, Study Director — Universidad Miguel Hernandez de Elche
Locations (1):
- University Miguel Hernández, Elche, Alicante, Spain